CLINICAL TRIAL: NCT05742204
Title: Identification and Functional Verification Study in Plasma Proteomic Biomarkers for Early Diagnosis of Lung Cancer
Brief Title: Plasma Proteomic Biomarkers for Early Diagnosis of Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1109
Record Dates: First submitted 2023-02-15; First posted 2023-02-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lung cancer group: Patients age over 18, with confirmed diagnosis of lung cancer.
  Interventions: Other: Plasma protein biomarker analysis
- Control group: Non-cancer patients including healthy volunteers, chronic inflammatory airway diseases such as chronic obstructive airway disease, asthma, and bronchiectasis, etc.
  Interventions: Other: Plasma protein biomarker analysis

INTERVENTIONS:
Other: Plasma protein biomarker analysis — Plasma samples from lung cancer patients were collected at the time of their diagnosis, prior to the initiation of treatment.We will use TMT-based proteomics approaches to analyze more than 2000 proteins in plasma samples from lung cancer patients .
  Groups: Lung cancer group
Other: Plasma protein biomarker analysis — Plasma samples of control subjects were collected.
  Groups: Control group

SUMMARY:
We will identify plasma proteomics biomarkers for early diagnosis of lung cancer.

DETAILED DESCRIPTION:
We will use TMT-based proteomics approaches to analyze more than 2000 proteins in plasma samples from lung cancer patients and controls. Artificial intelligent (AI) assisted proteomics classifier will be developed for early diagnosis of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* CT screening results showed that the size of pulmonary nodules was more than 5mm
* No treatment related to pulmonary nodules/lung cancer (including surgery, chemotherapy, radiotherapy, targeted therapy, immunotherapy, interventional therapy, etc.)
* Complete clinical and imaging data
* Chest CT/ low-dose spiral CT reports can be provided in the last 3 months
* Voluntarily sign informed consent

Exclusion Criteria:

* There is a history of tumor
* Clinically uncontrolled active infections, such as acute pneumonia, tuberculosis, etc.
* Received any treatment related to pulmonary nodules, such as antibiotics and hormones, in the past 4 weeks
* Complicated with other tumors and serious diseases of the heart, liver, kidney, brain, blood and other systems
* Participated in other clinical trials within the last 3 months
* Combined with liver and kidney insufficiency, hypoproteinemia and other diseases affecting protein content
* You are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study group: Patients with suspected or confirmed diagnosis of lung cancer. Control group: Non-cancer subjects including healthy volunteers, chronic inflammatory airway diseases such as chronic obstructive airway disease, asthma, and bronchiectasis, etc.
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Plasma proteomic biomarkers | 1 month after surgery
  Plasma proteomic biomarkers for detection of lung cancer
Model or classifier performance | 1 month after surgery
  Artificial intelligent (AI) assisted proteomics classifier will be developed for early diagnosis of lung cancer; and model or classifier performance including AUC, sensitivity, specificity, and accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Weilin Wang, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China, China

IPD SHARING:
Plan to Share IPD: Undecided